CLINICAL TRIAL: NCT00974688
Title: Optimizing Health Among Children With Congenital Heart Defects Through Rehabilitation Focused on Physical Activity Determinants
Brief Title: Optimizing Health Among Children With Congenital Heart Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1000012482
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Congenital Heart Defects
Keywords: Congenital; physical activity participation; Moderate-to-vigorous physical activity
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Behavioral: Information Intervention; Behavioral: Demonstration Intervention
- Group 2 (Active Comparator)
  Interventions: Behavioral: Information Intervention; Behavioral: Demonstration Intervention

INTERVENTIONS:
Behavioral: Information Intervention — The information intervention is designed to ensure that the parent(s) and child have a clear understanding of the range of physical activity opportunities that are appropriate and recommended for the child. The information intervention will be comprised of discussions and written information.
Behavioral: Demonstration Intervention — The demonstration intervention will be designed to demonstrate to the child and parent(s) specifically what the child is able to do in relation to fitness and motor skill activities. The demonstration intervention will consist of having the child complete a standardized exercise testing protocol on the treadmill, followed by discussions with the child and parent(s) to convey the results of the study testing of fitness and gross motor skill.

SUMMARY:
Quality of life and heart health are intimately connected to childhood physical activity participation (PAP). Physical activity is critical to childhood growth, development, learning, socialization, and quality of life and is an essential component of life-long heart health. Research by the investigators of this study and others has shown that low PAP levels are common among children with heart defects, and that these sedentary lifestyles are not related to exercise capacity, medical status or heart function.

DETAILED DESCRIPTION:
Therefore, we hypothesize that psychosocial factors are important determinants of PAP in this population. Our most recent research with children who have univentricular heart indicates that gross motor skill and psychosocial factors are significant correlates of PAP. Important psychosocial factors include self-efficacy for activity, uncertainty about activity, and inaccurate perceptions of the child's PAP level, options, and abilities. This study seeks to determine whether gross motor skill and psychosocial factors influence PAP among children with a broad spectrum of cardiac defects. It will also determine the optimal changes to clinical care needed to encourage children with heart defects to develop health-related active lifestyles.

We propose a prospective, randomized, cross-over preliminary clinical trial utilizing both quantitative and qualitative assessments. Through the cross-over design, each subject will complete both interventions (information, demonstration), with the order of intervention delivery randomly determined. Quantitative assessments will document moderate-to-vigorous physical activity (MVPA), gross motor skill, and health-related fitness. Qualitative assessments will evaluate parent/child anxiety about PAP and psychosocial factors influencing PAP. All factors will be assessed at each data collection point.

ELIGIBILITY:
Inclusion Criteria:

* Successful repair of one of the following congenital heart defects: transcatheter device closure of atrial septal defect (ASD), arterial switch repair of transposition of the great arteries (TGA), surgical repair of tetralogy of Fallot (TOF), or Fontan procedure for a functionally univentricular heart (UVH).
* At least one year after most recent open heart surgery.
* 4 to 11 years of age and attending elementary school at first study visit.

Exclusion Criteria:

* Identification of exercise contraindications/limitations by the responsible cardiologist.
* Other disabilities or medical conditions that may influence PAP. Children who achieve 90 minutes of MVPA on 5 or more days per week during the baseline assessment will be excluded from the intervention phase. The study interventions are not designed to increase MVPA among children who already achieve the Health Canada guidelines for PAP.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Difference in change of measured moderate-to-vigorous physical activity (MVPA) between groups | Baseline, 4, 8 and 12 month timepoints

SECONDARY OUTCOMES:
Gross motor skill | Baseline, 4, 8 and 12 month timepoints
Psychosocial variables | Baseline, 4, 8 and 12 month timepoints
Health-related fitness | Baseline, 4, 8 and 12 month timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Brain W McCrindle, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada